CLINICAL TRIAL: NCT02948101
Title: Pilot Study of the Pre-Conditioning Effects of Anti-Macrophage Therapy Using PD 0360324 in Recurrent Platinum-Resistant Epithelial Ovarian Cancer
Brief Title: PD 0360324 and Cyclophosphamide in Treating Patients With Recurrent High-Grade Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI's request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0053; NCI-2016-01928 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0053 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2016-10-25; First posted 2016-10-28 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (PD 0360324, cyclophosphamide) (Experimental): Patients receive anti-CSF1 monoclonal antibody anti-CSF1 monoclonal antibody PD 0360324 IV over 30 minutes on days 1, 8, 15, and 22. Starting on day 43, patients receive cyclophosphamide PO QD. Courses with cyclophosphamide repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Anti-CSF1 Monoclonal Antibody PD-0360324; Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Anti-CSF1 Monoclonal Antibody PD-0360324 — Given IV
  Other Names: Anti-M-CSF mAb PD-0360324; PD 0360324; PD 360324; PD-0360324; PD-360,324
Drug: Cyclophosphamide — Given PO
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies the side effects of PD 0360324 and cyclophosphamide and to see how well they work in treating patients with high-grade epithelial ovarian, primary peritoneal, or fallopian tube cancer that has come back after a period of improvement. Immunotherapy with monoclonal antibodies, such as PD 0360324, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Cyclophosphamide may stop the growth of disease by blocking the growth of new blood vessels necessary for tumor growth. Giving PD 0360324 and cyclophosphamide may work better in treating patients with high-grade epithelial ovarian, primary peritoneal, or fallopian tube cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the safety of anti-CSF1 monoclonal antibody PD-0360324 (PD 0360324) followed by cyclophosphamide in patients with epithelial ovarian, fallopian tube, and primary peritoneal cancers.

II. To examine the density of CD8+ T cells in tumor biopsies before and after PD 0360324.

SECONDARY OBJECTIVES:

I. To evaluate response rate and progression free survival associated with low dose oral cyclophosphamide after PD 0360324 treatment.

II. To evaluate M-CSF concentrations before and after treatment with PD 0360324 and during cyclophosphamide therapy.

TERTIARY OBJECTIVES:

I. To evaluate the immunologic effects of PD 0360324 on peripheral blood and ovarian cancer tissue.

II. To explore the relationships between drug concentration and immunologic biomarkers and response.

OUTLINE:

Patients receive anti-CSF1 monoclonal antibody PD 0360324 intravenously (IV) over 30 minutes on days 1, 8, 15, and 22. Starting on day 43, patients receive cyclophosphamide orally (PO) once daily (QD). Courses with cyclophosphamide repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 and 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histology showing recurrent high grade epithelial ovarian, peritoneal, or fallopian tube cancer
* Platinum resistant or refractory disease as defined by progression of disease on a platinum-containing regimen or recurrence of disease within 180 days of previous platinum treatment
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1; measurable disease is defined at least two lesions that can be accurately measured in at least one dimension (longest dimension to be recorded); each "target" lesion must be > 20 mm when measured by palpitation or >10 mm when measured by spiral computed tomography (CT), plain x-ray, magnetic resonance imaging (MRI), or positron emission tomography (PET)/CT; PET/CT will be acceptable at baseline if PET/CT was previously performed and available; imaging must be performed within -28 to -7 days of starting therapy; the target lesion must be distinct from other tumor areas selected for pre-treatment biopsies
* Subject must be willing to undergo protocol directed biopsies and blood draw for immune profiling
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of >= 4 months in the attending physician's estimation
* Estimated creatinine clearance > 40 mL/min by the Cockcroft-Gault formula
* White blood cell (WBC) >= 3.0 x 10^3/ul
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (> 1500 per mm^3)
* Platelet count >= 100 x 10^9/L (> 100,000 per mm^3)
* Hemoglobin >= 9.0 g/dL
* Female subjects must either be of non-reproductive potential (i.e., post-menopausal by history: >=60 years old and no menses for > 1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry
* Subject must be willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
* Signed informed consent for protocol PA13-0291

Exclusion Criteria:

* Absence of a biopsiable lesion as determined by radiologist
* Chemotherapy, hormonal, or biologic treatment for ovarian, fallopian tube, or primary peritoneal cancer in the last 21 days
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease >=5 years before the first dose of study drug and of low potential risk for recurrence;
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease; or
  * Adequately treated carcinoma in situ without evidence of disease, e.g. cervical cancer in situ
* Current or prior use of immunosuppressive medication within 21 days before the first dose of PD 0360324, with the exceptions of intranasal and inhaled corticosteroids and systemic corticosteroids at physiological doses (defined as not exceeding 10 mg/day of prednisone, or an equivalent dose of over corticosteroid)
* Prior immunotherapy with immune checkpoint inhibitors
* Any unresolved toxicity (> Common Terminology Criteria for Adverse Events [CTCAE] grade 1) from previous anti-cancer therapy with the exception of alopecia; subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripheral neuropathy)
* Subjects with an active infection requiring antibiotics or at an increased risk of latent infection that may affect safe study participation
* Subjects with existing periorbital edema
* Subjects with aspartate aminotransferase (AST) or alanine transaminase (ALT) >= 2 x upper limit of normal (ULN)
* Subjects with creatine kinase > ULN
* Subjects with clinically significant active ischemic heart disease, cardiac muscle disease (including cardiomyopathy or congestive heart failure) or myodegenerative disorders that may affect safe study participation
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days prior to study entry
* History of allergic or anaphylactic reaction to any therapeutic or diagnostic monoclonal antibody (IgG protein) or molecules made of components of monoclonal antibodies (e.g., Enbrel which is the Fc portion of an antibody or Lucentis which is a Fab)
* Pregnant or breastfeeding women or women of child-bearing potential who are not willing to use two highly effective methods of contraception (i.e., a hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence)
* Uncontrolled intercurrent illness including, but not limited to, bowel obstruction, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), tuberculosis, or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent, or undergo study procedures
* History of leptomeningeal carcinomatosis or brain metastasis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-31 (Estimated); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse effect | Up to 90 days
Density of CD8+ T cells in tumor biopsies | Up to 90 days
  Will be reported descriptively at each time point. Continuous measures will be presented with nonparametric methods such as median and interquartile range or boxplots, while correlations (Pearson's or Spearman's as indicated) will be calculated with other continuous measures. Scored or categorical measures will be tabulated.
Response rate | Up to 90 days
  Will be reported with a 95% confidence interval.
Progression-free survival | Up to 90 days
  Will be presented with a Kaplan-Meier curve.
Concentration-time data of PD 0360324 | Up to 90 days
  Will be summarized by descriptive statistics (n, mean, standard deviation, median, minimum, and maximum).

CONTACTS AND LOCATIONS:
Overall Officials: Amir Jazaeri, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org